CLINICAL TRIAL: NCT01386086
Title: Augmentation Therapy of Resistant Postpartum Depression With Aripiprazole
Brief Title: Aripiprazole and Resistant Postpartum Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Verinder Sharma, Psychiatrist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN138-623
Record Dates: First submitted 2011-04-21; First posted 2011-06-30 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Postpartum Depression
Keywords: Aripiprazole; adjunctive therapy; mood stabilizers; major depressive disorder; postpartum; Augmentation therapy; resistant
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder, Major | interventions — Aripiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Aripiprazole (Experimental): aripiprazole used adjunctively to antidepressants in patients with resistant postpartum depression
  Interventions: Drug: aripiprazole

INTERVENTIONS:
Drug: aripiprazole — The starting dose of aripiprazole will be 2 mg and the dose adjusted to a maximum of 15 daily

SUMMARY:
Currently there are no controlled data on the management of postpartum depression that fails to respond to adequate antidepressant therapy. The investigators recently reported that a large number of patients responded to the addition of atypical neuroleptics after having failed antidepressant trials. Aripiprazole used adjunctively to antidepressants is effective in patients with resistant depression but it has not been studied in patients with resistant postpartum depression. The investigators propose to conduct a 6 week open-label study to assess the effectiveness and tolerability of aripiprazole used adjunctively to antidepressants in patients with resistant postpartum depression.

ELIGIBILITY:
Inclusion Criteria:

* Euthyroid outpatients aged 18 to 45 years of age
* A DSM-IV diagnosis of major depressive disorder with episode onset within 3 months of delivery
* A 17-item HAM-D score of 18 or more
* Inadequate response to at least one antidepressant drug - defined as a <50% reduction in severity of depression for a duration of >6 weeks ( > than 8 weeks for fluoxetine), determined by the Massachusetts General Hospital Antidepressant Response Questionnaire. Patients having a score of 18 or more on the 17-item HAM-D will be eligible to participate in the study. The primary efficacy endpoint will be mean change in MADRS score, and the secondary endpoint will be mean change in the HAM-D score

  >For patients on psychotropic drugs (other than antidepressants) prior there will be a washout period of two weeks
* Ability to understand English and provide informed consent
* Women who delivered a healthy baby close to term (37-42 weeks)
* Use of adequate contraception > Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for at least 4 weeks after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.

WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or who is not post-menopausal.

Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicides) to prevent pregnancy, or who are practicing abstinence or where their partner is sterile (eg, vasectomy) should be considered to be of childbearing potential.

WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 7 days before the start of the investigational product.

A subject's male partner of fathering potential must use an adequate method of contraception to avoid conception throughout the study [and for at least 4 weeks after the last dose of study drug] to minimize the risk of pregnancy.

Exclusion Criteria:

* Women with onset of major depressive disorder during pregnancy
* Presence of another current Axis I disorder such as bipolar disorder, psychotic disorder or obsessive compulsive disorder or a history of psychosis or a history of post-partum mood disorder with psychotic features
* Presence of psychotic symptoms
* History of alcohol or substance abuse within the 12 months before screening
* Any Axis II diagnosis suggestive of likely non-compliance with study requirement or non-responsiveness to pharmacotherapy.
* Women receiving psychotherapy
* Women receiving psychotropic drugs not allowed in the study protocol
* Use of quinolone antibiotics such as ciprofloxacin
* Significant medical illness such as end stage renal disease, uncontrolled narrow angle glaucoma and liver disease
* Women considered at high risk for suicide-those that are actively suicidal or have a score of ≥ 3 on item #3 on the 17-item HAMD; or women who, in the opinion of the Investigator, are deemed to be at risk of causing harm to the baby
* Women who are nursing/breastfeeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | 6 weeks
  To assess the effectiveness of the addition of aripiprazole in the treatment of resistant postpartum depression as measured by the change in mean scores on the Montgomery Asberg Depression Rating Scale between baseline and the study termination endpoint.

SECONDARY OUTCOMES:
Udvalg for Kliniske Undersogelser Scale | 6 weeks
  To assess the tolerability of aripirazole in women with resistant postpartum depression as assessed by the Udvalg for Kliniske Undersogelser Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Verinder Sharma, MBBS, Principal Investigator — Western University, Canada
Locations (1):
- Regional Mental Health Care, London, Ontario, Canada